CLINICAL TRIAL: NCT06787118
Title: Randomized, Double-blind, Placebo-controlled, 2x2 Cross Over Study Assessing the Efficacy and Safety of cANnabidiol Oral Solution for Joint Pain of Adjuvant enDOcrine theRApy in Patients With Early Breast Cancer
Brief Title: Study Assessing the Efficacy and Safety of cANnabidiol Oral Solution for Joint Pain of Adjuvant enDOcrine theRApy in Patients With Early Breast Cancer
Acronym: PANDORA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023-505380-36-01; 2021/3373 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III; HR+ Breast Cancer; AI-related Musculoskeletal Pain
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (CBD then Placebo) (Experimental): 12 weeks CBD-oral solution 2.5 mg/kg x 2/day followed by 12 weeks placebo. A 1-week off-therapy period (wash out) +/-2 days will be performed between study periods.
  Interventions: Drug: CBD oil; Drug: Placebo
- Arm 2 (Placebo then CBD) (Experimental): 12 weeks Placebo followed by 12 weeks CBD-oral solution 2.5 mg/kg x 2/day (5 mg/kg/day).
  A 1-week off-therapy period (wash out) +/-2 days will be performed between study periods.
  Interventions: Drug: CBD oil; Drug: Placebo

INTERVENTIONS:
Drug: CBD oil — Patients will receive CBD-oral solution 2.5 mg/kg PO BID for a total of 12 weeks.
Drug: Placebo — Patients will receive placebo for a total of 12 weeks.

SUMMARY:
Phase III, single-center, randomized, double-blind, placebo-controlled, 2x2 cross- over study, assessing the efficacy of CBD in patients with early HR+ BC, presenting aromatase inhibitor-related musculoskeletal pain

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria:

1. Patient must understand, sign and date the written informed consent form (ICF) prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedure as per protocol.
2. Patient must be affiliated to a social security system or beneficiary of the same.
3. Patient is ≥ 18 years-old at the time of study inclusion
4. Patient has histologically confirmed invasive Stage I, II, III breast cancer.
5. Patient has breast cancer that is positive for ER and/or PgR (nuclear staining of any intensity ≥ 10%)
6. Patients should be taking a standard dose of one of the three approved AIs (i.e., anastrozole, exemestane, or letrozole) for at least 21 days, and not more than 36 months before trial registration; premenopausal patients are eligible if they are receiving AIs and ovarian function suppression (LHRH agonist).
7. If indicated, patient has completed adjuvant and/or neoadjuvant chemotherapy according to the institutional guidelines, prior to randomization.
8. If indicated, patient has completed adjuvant radiotherapy according to the institutional guidelines, prior to randomization.
9. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
10. Patients should report an Interference pain score of ≥ 4 out of 10 on the Brief Pain Inventory (BPI, Appendix 2) within 7 days before registration.
11. Patient must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other trial procedures.
12. Women of childbearing potential (CBP), defined as all women physiologically capable of becoming pregnant, must have confirmed negative urine or serum pregnancy test (for β- hCG) within 14 days of randomization.
13. Women of CBP, defined as all women physiologically capable of becoming pregnant, must be willing to use highly effective methods of contraception. It is recommended that sexually active males use a condom during intercourse and it is strongly advised that they do not father a child in this period (a condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via seminal fluid). In all patients, contraception must continue during the trial treatment and for 3 months after stopping it, due to AI treatment. For women, highly effective contraception methods include:

    1. Total abstinence (when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception;
    2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks before taking trial treatment. In case of bilateral oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment;
    3. Placement of an intrauterine device (IUD). Notes:

       * Use of oral (estrogen and progesterone), transdermal, injected or implanted hormonal methods of contraception (as well as hormonal replacement therapy) is not allowed in this trial.
       * Women are considered of CBP unless: they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks ago.

    Specific inclusion criteria for CBD use:
14. Patient has adequate bone marrow and organ function as defined by the following local laboratory values:

    1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
    2. Platelets ≥ 100 × 109/L
    3. Hemoglobin ≥ 9.0 g/dL
    4. Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min by a Cockcroft-Gault formula.
    5. Alanine transaminase (ALT) ≤ 1.5 × Upper Limit Normal (ULN)
    6. Aspartate transaminase (AST) ≤ 1.5 × ULN
    7. Total serum bilirubin ≤ ULN; or total bilirubin ≤ 3.0 × ULN with direct bilirubin ≤ 1.5 × ULN in patients with well documented Gilbert's Syndrome
    8. International normalized ratio (INR) ≤ 1.5 (unless the patient is receiving anticoagulants and the INR is within the therapeutic range of intended use for that anticoagulant within 7 days prior to randomization).
    9. Patient must have the following laboratory values within normal limits or corrected to within normal limits with supplements (the local laboratory value should be documented within normal limits after the correction) before randomization:

       * Sodium
       * Potassium
       * Phosphorus
       * Magnesium
       * Total Calcium
15. Standard 12-lead ECG values defined as the mean of the triplicate ECGs as locally assessed:

    1. QTcF interval (using Fridericia's correction) at screening < 450 msec
    2. Mean resting heart rate 50-90 bpm (determined from the ECG)

Exclusion Criteria:

General exclusion criteria:

1. Patient with distant metastases of breast cancer beyond regional lymph nodes (M1 disease according to AJCC 8th edition).
2. Patient has not recovered from clinical and laboratory acute toxicities of chemotherapy, radiotherapy and/or surgery (i.e. patient has toxicities attributed to prior anti-neoplastic therapy NCI CTCAE version 5.0 grade ≥1 at day of randomization, excluding alopecia and amenorrhea)
3. Patient has a concurrent invasive malignancy or a prior invasive malignancy whose treatment was completed within 2 years before ICF signature. Note: Patients with prior or concurrent in situ malignancies are eligible provided that adequate curative treatment is completed prior to randomization
4. Patient has previous history of bone fracture or surgery of the affected knees, hands or both within 6 months prior to enrolment or known rheumatologic diseases;
5. Patient has received opioids analgesics, systemic NSAIDs, topical analgesics, oral, intra-articular or intramuscular corticosteroids for treatment of joint pain or joint stiffness within 28 days prior registration;
6. Patient has active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
7. Patients with moderate (Child-Pugh B) hepatic impairment or severe (Child-Pugh C) hepatic impairment.
8. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the oral trial treatments (e.g. uncontrolled ulcerative diseases, uncontrolled nausea, vomiting or diarrhea, malabsorption syndrome, or small bowel resection).
9. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the Investigators judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical trial or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, liver cirrhosis or any other significant liver disease, active untreated or uncontrolled fungal, bacterial or viral infections, active infection requiring systemic anti-bacterial therapy, etc.) or limit life expectancy to ≤5 years.
10. Participation in a prior interventional study and received trial treatment with an investigational product (or used an investigational device) within 30 days prior to randomization or within 5 half-lives of the investigational product, whichever is longer.
11. Pregnant or breast-feeding (lactating) women or women who plan to become pregnant or breastfeed during the trial.
12. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or under justice protection or under curatorship or unable of giving his consent

    Specific exclusion criteria for CBD use:
13. Patient with a known hypersensitivity to CBD or any of the excipients of CBD
14. Previous serious adverse reaction to any cannabinoid product such as cannabinoid related psychosis, panic attack or delirium.
15. Recreational or medicinal cannabis or synthetic cannabinoid based medications (including Sativex®) within 2 weeks before study entry
16. Patient has previous or active psychological, psychiatric or central nervous system disorders, including epilepsy; schizophrenia or any other psychosis, severe borderline personality, patient with significant suicidal ideation.
17. Patient takes drugs as clobazam, valproate, or levodopa;
18. Patient has previous history of substance abuse or dependence to alcohol, opioids, amphetamines, benzodiazepines and other illicit stimulants.
19. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:

    1. History of documented myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to trial entry
    2. Documented cardiomyopathy
    3. Prior history of LVEF <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) which did not recover before study entry
    4. Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

       * Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia
       * Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause TdP that cannot be discontinued or replaced by safe alternative medication (e.g. within 5 half-lives or 7 days prior to starting trial treatment)
       * Inability to determine the QTcF interval
    5. Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade Atrioventricular (AV) block (e.g. bifascicular block, Mobitz type II and third degree AV block)
    6. Uncontrolled arterial hypertension with systolic blood pressure (SBP) > 160 mmHg

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory - Short Form (BPI-SF) Interference score. | Baseline, 4 weeks, 12 weeks, 13 weeks, 17 weeks, 25 weeks, 37 weeks after starting treatment.
  The BPI is a 14-item questionnaire that asks patients to rate pain over the last 24 hours and the degree to which it interfered with activities on a 0-10 scale, where higher scores indicate more pain.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis scale (WOMAC). | Baseline, 4 weeks, 12 weeks, 13 weeks, 17 weeks, 25 weeks, 37 weeks after starting treatment.
  This is a 24-item questionnaire that is used to assess pain, stiffness, and functioning in the knees and hips during the past week.
  The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores.[1]
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
EORTC QLQ-C30 | Baseline, 4 weeks, 12 weeks, 13 weeks, 17 weeks, 25 weeks, 37 weeks after starting treatment.
  The EORTC Quality of Life Questionnaire-C30 (EORTC QLQ-C30) contains 30 questions and assesses the quality of life of oncological patients multidimensionally over 10 subscales. All sub-scales and the 6 individual items have a score range from 0 to 100 points. A higher score represents better function and a higher quality of life. In the symptom subscale, however, a higher score represents a higher level of symptoms or problems.
EORTC QLQ-BR45. | Baseline, 4 weeks, 12 weeks, 13 weeks, 17 weeks, 25 weeks, 37 weeks after starting treatment.
  The QLQ-BR45 is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30. The QLQ-BR45 incorporates nine multi-item scales to assess body image, sexual functioning, breast satisfaction, systemic therapy side effects, arm symptoms, breast symptoms, endocrine therapy symptoms, skin mucosis symptoms, endocrine sexual symptoms. In addition, single items assess sexual enjoyment, future perspective and being upset by hair loss. All of the scales and single item measures range in score from 0 to 100. A high score for the functional scales and functional single items represents a high/healthy level of functioning, whereas a high score for the symptom scales and symptom item represents a high level of symptomatology or problems.
EORTC QLQ-FA12. | Baseline, 4 weeks, 12 weeks, 13 weeks, 17 weeks, 25 weeks, 37 weeks after starting treatment.
  The FA12 is the new fatigue module designed to complement the EORTC QLQ-C30. It consists of 12 items, with four response categories for each item, coded with values from 1 to 4. In accordance with the scales of the EORTC QLQ-C30, the FA12 scores are transformed to the range 0-100, with higher levels indicating greater degrees of fatigue.
Hospital Anxiety and Depression Scale (HADS). | Baseline, 4 weeks, 12 weeks, 13 weeks, 17 weeks, 25 weeks, 37 weeks after starting treatment.
  HADS is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.
Medication intake survey (MIS). | Baseline, 4 weeks, 12 weeks, 13 weeks, 17 weeks, 25 weeks, 37 weeks after starting treatment.
  A 10-item survey, representing a French validated self-report instrument measuring key adherence properties. Taking adherence is computed over 1 week, 4 weeks and 4 months. A high score represents a high level of adherence
Adherence | Baseline, 4 weeks, 12 weeks, 13 weeks, 17 weeks, 25 weeks, 37 weeks after starting treatment.
  Patient's self-reporting through the questionnaire MIS
Domain-Specific Risk-Taking (DOSPERT) scale. | Baseline.
  The DOSPERT is a risk-taking scale of the 30-item evaluates behavioral intentions, that is, the likelihood with which respondents might engage in risky behaviors originating from five domains of life (ethical, financial, health/safety, social, and recreational risks) using a 7-point rating scale ranging from 1 (Extremely Unlikely) to 7 (Extremely Likely). Higher scores suggesting perceptions of greater risk in the domain of the subscale.
Number of side effects measured by CTCAE V.5. | Baseline, 4 weeks, 12 weeks, 13 weeks, 17 weeks, 25 weeks, 37 weeks after starting treatment.
  An adverse event (AE) is defined as any untoward medical occurrence, in a patient or clinical trial subject treated by a medicinal product and which does not necessarily have a causal relationship with this treatment. The AE collected will be particularly focused on nausea, diarrhea or constipation, cognitive dysfunction, nervous system and psychiatric side effects, drug consumption and hospitalizations associated with nervous system and psychiatric disorders.
Cannabis Abuse Screening Test (CAST). | Baseline, 4 weeks, 12 weeks, 13 weeks, 17 weeks, 25 weeks, 37 weeks after starting treatment.
  The CAST scale is a 6-item scale evaluating cannabis abuse among adolescents and young adults in general population surveys designed at the French Monitoring Center for Drug and Drug addictions (OFDT). A score of less than 3 indicates no addiction risk. A score of 3 or less than 7 indicates low addiction risk, and a score of 7 or above indicates high addiction risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: In 2018, Little Green Pharma pioneered the Australian medical cannabis market and were able to launch Australia's first locally grown cannabis medicine. — https://www.littlegreenpharma.com/au/